CLINICAL TRIAL: NCT07398833
Title: Modulation of Working Memory by an Alternating Magnetic Field in Humans
Acronym: MEMOCHAM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Beau Soleil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2025-A00296-43
Record Dates: First submitted 2025-12-08; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Healthy
MeSH Terms: interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 40 Hz tACS stimulation (Experimental)
  Interventions: Other: Electrical stimulation
- 60 Hz tACS stimulation (Experimental)
  Interventions: Other: Electrical stimulation
- 40 Hz tAMS stimulation (Experimental)
  Interventions: Other: Magnetic stimulation
- 60 Hz tAMS stimulation (Experimental)
  Interventions: Other: Magnetic stimulation
- No stimulation (Sham Comparator)
  Interventions: Other: No stimulation

INTERVENTIONS:
Other: Electrical stimulation — The experimental session lasts 2 hours and 30 minutes and includes four phases: Time 0, dedicated to training and adjustment of task difficulty, followed by Time 1, Time 2, and Time 3, corresponding respectively to assessments of working memory performance before, during, and after exposure to stimulation. Each phase includes blocks of the Sternberg task, for a total of 180 trials per session. Each block lasts 10 minutes.
  Arms: 40 Hz tACS stimulation; 60 Hz tACS stimulation
Other: Magnetic stimulation — The experimental session lasts 2 hours and 30 minutes and includes four time points: Time 0, dedicated to training and adjustment of task difficulty, followed by Time 1, Time 2, and Time 3, corresponding respectively to assessments of working memory performance before, during, and after exposure to stimulation. Each time point includes blocks of the Sternberg task, for a total of 180 trials per session. Each block lasts 10 minutes.
  Arms: 40 Hz tAMS stimulation; 60 Hz tAMS stimulation
Other: No stimulation — The experimental session lasts 2 hours and 30 minutes and includes four time points: Time 0, dedicated to training and adjustment of task difficulty, followed by Time 1, Time 2, and Time 3, corresponding respectively to assessments of working memory performance before, during, and after exposure to sham stimulation. Each time point includes blocks of the Sternberg task, for a total of 180 trials per session. Each block lasts 10 minutes.
  Arms: No stimulation

SUMMARY:
Many studies have examined the effects of transcranial alternating current stimulation (tACS) on working memory, showing that low-intensity stimulation can enhance cognitive performance by modulating neuronal activity, particularly in the frontal cortex and the parietal lobule. Specific frequencies, such as the gamma frequency, have demonstrated beneficial effects on memory under high cognitive load. However, tACS has technical limitations, including uncomfortable sensations and uneven diffusion of electrical currents within the brain, which restrict its effectiveness in deeper brain regions.

Transcranial alternating magnetic stimulation (tAMS) is emerging as a potentially more precise and comfortable method. Unlike tACS, tAMS uses magnetic fields that penetrate more deeply into the brain and provide a more homogeneous distribution of induced electrical currents, allowing for more targeted stimulation. This study compares the effects of tACS and tAMS on working memory, with the hypothesis that tAMS will offer additional advantages in terms of comfort and efficacy. Cognitive performance will be assessed using working memory tasks, along with EEG signals to analyze neuronal modulations. The objective is to demonstrate that tAMS more effectively reaches deep brain regions and improves cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* Written, voluntary, and informed consent to participate in the study
* Fluent French speaker (task instructions are provided in French)
* Normal or corrected-to-normal vision using contact lenses only

Non inclusion Criteria:

* Individuals deprived of liberty by law
* Individuals under legal guardianship or curatorship
* Pregnant or breastfeeding women
* Presence of metallic implants in the head, implanted electronic devices, or any other metallic object that cannot be removed for the experiment (e.g. dental fillings)
* History of neurological or psychiatric disorders according to the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition)
* History of pathology or chronic disease affecting memory or attention
* Drug or alcohol consumption within the previous 24 hours

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Sternberg task | Baseline (Day 1, before exposure), periprocedural (Day 1, during exposure), and post-intervention (Day 1, immediately after exposure)
  During each trial, participants memorize a sequence of eight letters presented sequentially. They are then shown a probe letter displayed in blue and must indicate whether this letter was part of the memorized sequence. Participant performance will be evaluated based on two behavioral measures: accuracy (proportions of correct and incorrect responses) and reaction time in milliseconds.

SECONDARY OUTCOMES:
EEG Power Outcomes | Baseline (Day 1, before exposure), periprocedural (Day 1, during exposure), and post-intervention (Day 1, immediately after exposure)
  Absolute power of EEG frequency bands will be measured using power spectral density analysis to quantify the energy within each frequency band associated with working memory.
EEG Power Outcomes | Baseline (Day 1, before exposure), periprocedural (Day 1, during exposure), and post-intervention (Day 1, immediately after exposure)
  Relative power of EEG frequency bands will be calculated as the proportion of power in each frequency band relative to the total EEG signal power.
EEG Power Outcomes | Baseline (Day 1, before exposure), periprocedural (Day 1, during exposure), and post-intervention (Day 1, immediately after exposure)
  Mean frequency of the EEG signal will be calculated from the power spectral density to characterize frequency distribution related to working memory processes.
EEG Power Outcomes | Baseline (Day 1, before exposure), periprocedural (Day 1, during exposure), and post-intervention (Day 1, immediately after exposure)
  Median frequency of the EEG signal will be derived from the power spectral density as an indicator of the central tendency of EEG frequency content.
EEG Power Outcomes | Baseline (Day 1, before exposure), periprocedural (Day 1, during exposure), and post-intervention (Day 1, immediately after exposure)
  Peak power frequency of the EEG signal will be identified as the frequency at which maximum power occurs.
EEG Signal Regularity Outcomes (RQA) | Baseline (Day 1, before exposure), periprocedural (Day 1, during exposure), and post-intervention (Day 1, immediately after exposure)
  Recurrence rate derived from recurrence quantification analysis will be used to quantify the proportion of recurrent patterns in the EEG signal.
EEG Signal Regularity Outcomes (RQA) | Baseline (Day 1, before exposure), periprocedural (Day 1, during exposure), and post-intervention (Day 1, immediately after exposure)
  Determinism derived from recurrence quantification analysis will be used to assess the temporal organization and regularity of EEG signal dynamics.
Neuropsychological data | Baseline (Day 1, before exposure)
  Score from the Multidimensional Fatigue Inventory (MFI-20) will be used to assess fatigue.
  The Multidimensional Fatigue Inventory is a self-reported questionnaire with total scores ranging from 20 to 100. Higher scores reflect higher levels of fatigue.
Neuropsychological data | Baseline (Day 1, before exposure)
  Score from the State-Trait Anxiety Inventory (STAI) will be used to assess anxiety.
  The State-Trait Anxiety Inventory is a self-reported questionnaire with scores ranging from 20 to 80. Higher scores reflect higher levels of anxiety.